CLINICAL TRIAL: NCT00004315
Title: Phase II Pilot Study to Compare the Bioavailability of Buffered, Enteric-Coated Ursodiol With Unmodified Ursodiol for Chronic Cholestatic Liver Disease and Cystic Fibrosis-Associated Liver Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Purpose: Treatment
Other Study IDs: 199/11827; UCMC-CHMC-915717
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-04

CONDITIONS: Cystic Fibrosis; Gastrointestinal Diseases; Cholestasis
Keywords: cardiovascular and respiratory diseases; cholestasis; cystic fibrosis; gastrointestinal disorders; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Gastrointestinal Diseases; Cholestasis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases | interventions — Ursodeoxycholic Acid

INTERVENTIONS:
Drug: ursodiol

SUMMARY:
OBJECTIVES: I. Compare the bioavailability of polymer-coated and buffered ursodiol (ursodeoxycholic acid) to unmodified ursodiol in patients with cystic fibrosis-associated liver disease or chronic cholestatic liver disease.

II. Compare the differences in pruritus, weight gain, and liver function for both treatments.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are sequentially treated with 2 formulations of ursodeoxycholic acid: unmodified ursodiol (Actigall) and buffered, enteric-coated ursodiol (Ursocarb). There is a 24-hour washout between each 4-week course of therapy.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Chronic cholestatic liver disease

Cystic fibrosis-associated liver disease

--Prior/Concurrent Therapy--

Usual and customary diet maintained throughout study, e.g., medium-chain triglyceride oil

--Patient Characteristics--

Pulmonary: No serious respiratory deficiency

No acute illness

No inability to swallow

No fertile women

Min Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1995-11

CONTACTS AND LOCATIONS:
Overall Officials: William Balistreri, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio, United States